CLINICAL TRIAL: NCT04846686
Title: Placental Expression of EG-VEGF and Its PROKR1 and PROKR2 Receptors in Preeclampsia Patients.
Acronym: PRE-EVE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Commissariat A L'energie Atomique (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRBN622021/CHUSTE
Record Dates: First submitted 2021-04-13; First posted 2021-04-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; EG-VEGF; Prokineticin; cesarean; placenta pathological examination; pregnancy; PROK1 receptor; PROKR2 receptor
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — placental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- preeclampsia group: 25 patients with a diagnostic of preeclampsia, having undergone a placental pathological examination and having given birth by cesarean section. A cross-referencing of data with programme for medicalization of information systems (PMSI) will be realized.
  Placenta pathological examination will be performed.
  Interventions: Biological: Placenta pathological examination
- control group: 10 patients who had a normal pregnancy, having undergone a placental pathological examination and having given birth by cesarean section. A cross-referencing of data with PMSI will be realized.
  Placenta pathological examination will be performed.
  Interventions: Biological: Placenta pathological examination

INTERVENTIONS:
Biological: Placenta pathological examination — a placenta pathological examination will be analyzed to examine quantification of EG-VEGF, PROKR1 and PROKR2 receptors.

SUMMARY:
The pathophysiology of preeclampsia (PE) is thought to be endothelial dysfunction responsible for the maternal signs of de novo hypertension and proteinuria after 20 weeks. Current concepts suggest that the pathophysiology of preeclampsia and intrauterine growth retardation results from an imbalance of angiogenic factors.

A new angiogenic factor EG-VEGF (Endocrine Gland- Derived Vascular Endothelial Growth Factor) also known as Prokineticin 1 (PROK1) appears to be emerging in the pathophysiology of PE. EG-VEGF is a circulating factor which belongs to the family of prokinetics. Dr Alfaidy's MAB2 team at the Cancer and Infections Biology Laboratory (U1292 Biosanté INSERM / UGA / CEA, CEA Grenoble) demonstrated its key role in the control of key processes in placental development and provided evidence through the development of an animal model of preeclampsia. EG -VEGF is directly involved in the development of Pre-Eclampsia. Few studies have evaluated the expression of EG-VEGF in the human placenta.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have given birth by cesarean section at the maternity University Hospital Saint Etienne and all underwent a placenta pathological examination at the Saint Etienne University Hospital.
* For the pre-eclampsia group: patient with a diagnosis of pre-eclampsia
* For the control group: patient who had a normal pregnancy

Exclusion Criteria:

* Patient who gave birth naturally
* Underage patients or under guardianship
* Patients who do not speak or read French
* Childbirth under X

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who have given birth by cesarean section at the maternity University Hospital Saint Etienne and all underwent a placenta pathological examination at the Saint Etienne University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Immuno-localization of EG-VEGF staining (ImageJ®) by immunohistochemistry | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).
Quantification of EG-VEGF staining (ImageJ®) by immunohistochemistry | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).

SECONDARY OUTCOMES:
Immuno-localization of the staining of PROKR1 (ImageJ®) by immunohistochemistry | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).
Quantification of the staining of PROKR1 (ImageJ®) by immunohistochemistry | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).
Immuno-localization of the staining of PROKR2 (ImageJ®) by immunohistochemistry | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).
Quantification of the staining of PROKR2 (ImageJ®) by immunohistochemistry Measure by placenta pathological examination (immunohistochemistry technical). | At delivery
  Measured by placenta pathological examination (immunohistochemistry technical).
Presence of at least one chronic maternal pathologies describe below | At delivery
  diabetes, hypertension, kidney disease, Systemic Lupus Erythematosus (SLE), antiphospholipid syndrome
Obstetric history | At delivery
  Pre-Eclampsia (PE) and intra uterine growth retardation (IUGR), term of onset and severity of Pre-Eclampsia (PE)
Presence of an anticoagulant treatment | At delivery
  treatment by aspirin or Heparin or low molecular weight heparins (LMWH)

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine BARJAT, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No